CLINICAL TRIAL: NCT01745679
Title: Therapeutic Monitoring of Ceftriaxone, Prescribed at High Doses, in the Treatment of Meningitis and Others Neurological Infections.
Brief Title: Pharmacological Study of High Doses of Ceftriaxone in Meningitidis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RC12_0171
Record Dates: First submitted 2012-12-04; First posted 2012-12-10 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Meningitis; Neurological Infections
Keywords: Ceftriaxone; Adverse drug effects; Therapeutic monitoring; Meningitis
MeSH Terms: conditions — Meningitis; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ceftriaxone treatment (Experimental): ceftriaxone will be administered à high dose : > or equal to 75mg/kg/day or 4 gr/day
  Interventions: Drug: Ceftriaxone treatment

INTERVENTIONS:
Drug: Ceftriaxone treatment — ceftriaxone will be administered à high dose : > or equal to 75mg/kg/day or 4 gr/day

SUMMARY:
The aim of the study is to describe the concentrations of Ceftriaxone at the steady state, in patients treated for meningitis, to determine pharmacokinetic parameters at high dose in this population. Additionally, we aimed to detect adverse effect, especially neurological trouble related to Ceftriaxone toxicity.

DETAILED DESCRIPTION:
Day 0 : onset of treatment by Ceftriaxone, following usual therapeutic process (French Guideline) From Day 0 to Day 4 : inclusion, clinical and biological data collection, electroencephalogram at baseline.

Two samples for ceftriaxone concentration monitoring :

* Trough concentration of ceftriaxone at steady state
* A random sample (population PK) At the end of ceftriaxone treatment : assessment of tolerance and efficacy of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adults patients,
* age equal or above 18
* Patients with Community or surgical acquired neurological infections, meningitis and others
* Prescription of ceftriaxone >75mg/kg/d or >4g/d -
* Subjects affiliated to French health insurance (social security)
* Informed consent form signed

Exclusion Criteria:

- Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
plasmatic concentration of ceftriaxone, measured at the steady state (after 48 hours of treatment at least). | after at least 48 hours of ceftriaxone treatment

SECONDARY OUTCOMES:
Neurological troubles | participants will be followed for the duration of ceftriaxone treatment, an expected average of two weeks
  Neurological troubles explored by electroencephalogram aiming to diagnose epileptic syndrome.
clinical evolution | participants will be followed for the duration of ceftriaxone treatment, an expected average of 2 weeks
  Time of return to apyrexia, health complications and lenght of hospital stay will be registered.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Tours universitary hospital, Tours, France
  - Nantes Universitary Hospital, Nantes, Loire Atlantique
  - Angers Universitary Hospital, Angers
  - La Roche/Yon hospital, La Roche/Yon
  - Poitiers Universitary hospital, Poitiers
  - Rennes Universitary hospital, Rennes
  - St Nazaire hospital, Saint-Nazaire

REFERENCES:
- [Derived] Gregoire M, Dailly E, Le Turnier P, Garot D, Guimard T, Bernard L, Tattevin P, Vandamme YM, Hoff J, Lemaitre F, Verdier MC, Deslandes G, Bellouard R, Sebille V, Chiffoleau A, Boutoille D, Navas D, Asseray N. High-Dose Ceftriaxone for Bacterial Meningitis and Optimization of Administration Scheme Based on Nomogram. Antimicrob Agents Chemother. 2019 Aug 23;63(9):e00634-19. doi: 10.1128/AAC.00634-19. Print 2019 Sep. PMID 31235630